CLINICAL TRIAL: NCT06073665
Title: Levothyroxine Dosing in Older Individuals
Brief Title: Dosing of LT4 in Older Individuals
Acronym: DOT4
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Anne Cappola, MD, Professor of Medicine, Division of Endocrinology, Diabetes and Metabolism, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01AG081698-01 (NIH); R01AG081698 (NIH)
Record Dates: First submitted 2023-09-22; First posted 2023-10-10 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Hypothyroidism
Keywords: Levothyroxine Dosing
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Intervention Model Description: randomized, parallel, double-blind clinical trial of two 6-month dosing strategies of levothyroxine (LT4)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: overencapsulated levothyroxine doses will be provided by the investigational drug pharmacy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lower TSH Group (Active Comparator): Target TSH level of 0.5-2.0 mU/L
  Interventions: Drug: Levothyroxine Sodium
- Higher TSH group (Experimental): Target TSH level of 5.5-7.0 mU/L
  Interventions: Drug: Levothyroxine Sodium

INTERVENTIONS:
Drug: Levothyroxine Sodium — Levothyroxine dose will depend on dose at baseline and randomization group

SUMMARY:
Our overall goal is to determine the clinical consequences of allowing greater flexibility in LT4 dosing in older individuals who take LT4.

DETAILED DESCRIPTION:
Investigators will perform a randomized, parallel, double-blind clinical trial of two 6-month dosing strategies of levothyroxine (LT4) in patients aged 65 years and older who are already taking a stable dose of at least 1.2 mcg/kg/day of LT4 therapy, one to maintain a target thyroid stimulating hormone (TSH) level of 0.5-2.0 mU/L (lower TSH group) and another of a lower levothyroxine dose to achieve a target TSH of 5.5-7.0 mU/L (higher TSH group). Investigators will assess the effects of levothyroxine therapy at two different TSH targets on symptoms of hypothyroidism, mood, sleep, measures of memory and executive function, weight, lipids, and a marker of bone turnover.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, community dwelling, aged 65 years or older
4. Diagnosed with hypothyroidism of any etiology for at least 6 months, taking 75-200 mcg per day LT4 and a minimum of 1.2 mcg/kg/day with no dose adjustment since the last TSH test.
5. Ability to take oral medication and be willing to adhere to the medication regimen

Exclusion Criteria:

1. Hypopituitarism
2. History of thyroid cancer requiring suppression of TSH secretion
3. Current use of liothyronine (LT3), thyroid extracts, Tirosint liquid or capsules, and medications that interfere with thyroid function or thyroid function tests
4. GFR <30 ml/min/1.73 m2 within the prior 12 months
5. Unable to understand and comply with study requirements, as assessed by study staff and the PI, will be excluded.
6. Other conditions which, in the opinion of the investigators, would prevent them from participating in the full duration of the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Thyroid-Related Quality of Life Patient-Reported Outcome Quality of Life scale | 6 months
  22 items, scored 0-100, higher scores indicate worse status

SECONDARY OUTCOMES:
Thyroid-Related Quality of Life Patient-Reported Outcome Hypothyroidism subscale b. ThyPRO "Tiredness" subscale c. Thyroid Symptoms Questionnaire (TSQ) | 6 months
  4 items, scored 0-100, higher scores indicate worse status
NIH Toolbox Fluid Cognition Composite Score | 6 months
  Adjusted scale score, based around median of 100, higher scores indicated higher function
Geriatric Depression Scale | 6 months
  30 items, higher scores indicate more depressive symptoms
Pittsburgh Sleep Quality Index | 6 months
  19 items, range of 0-21, higher scores indicate worse sleep
Weight | 6 months
  kilograms
LDL cholesterol | 6 months
  blood test, g/dL
Satisfaction with randomized status | 6 months
  Participants will be asked if they can guess their randomization status and satisfaction with randomization status
Beck Anxiety Inventory | 6 months
  Beck Anxiety Inventory, 21 items, range 0-63, higher scores indicate more anxiety
Serum c-telopeptide (CTX) | 6 months
  Blood test, pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Anne R. Cappola, M.D., Sc.M., Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Medicine, Smilow Translational Research Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No